CLINICAL TRIAL: NCT01218230
Title: A Clinical Trial to Study the Efficacy and Safety of Intravitreal Pegaptanib in Treatment of Choroidal Neovascularisation Secondary to Pathologic Myopia
Brief Title: Intravitreal Pegaptanib in Treatment of Choroidal Neovascularisation Secondary to Pathologic Myopia
Acronym: INGECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding did not come through as the product was sold to another company.
Sponsor: L.V. Prasad Eye Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Raja Narayanan, Head of Clinical Research, L.V. Prasad Eye Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEC08205
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Myopic Choroidal Neovascular Membrane
Keywords: Pegaptanib, myopic CNVM, intravitreal anti-VEGF
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Pegaptanib (Active Comparator)
  Interventions: Drug: Intravitreal Pegaptanib

INTERVENTIONS:
Drug: Intravitreal Pegaptanib — Intravitreal pegaptanib, 0.3 mg, every 6 weeks for 3 injections and then PRN.
  Other Names: Macugen

SUMMARY:
Intravitreal pegaptanib for treatment of choroidal neovascularisation secondary to pathologic myopia

DETAILED DESCRIPTION:
This is a Prospective Interventional, non-comparative study in 20 consecutive patients who will be selected from the outpatient services. After taking an informed consent, the patients will be given intravitreal Pegaptanib 0.3 mg every 6 weeks for 3 procedure of injection. Thereafter, patients will continue to be examined every 6 weeks (± 2 weeks) and of may receive additional injections as needed based on the presence of one or more re-treatment criteria (please see below). Final assessment will be done at 54 weeks and all the baseline investigations will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Should be willing to participate in the trial.
2. Age less than 55 years.
3. Best corrected visual acuity (BCVA) score of at least 5 letters (20/200), as assessed by ETDRS chart.
4. Myopia of ≥ 6 Diopters.
5. Fluorescein angiographic documentation of CNV.

Exclusion Criteria:

1. Ocular causes, or other ocular disorders leading to vision loss.
2. Maculopathy not related to pathologic myopia.
3. Pregnancy, lactation.
4. Not willing to provide an informed consent.
5. History of previous macular laser including PDT.
6. Other forms of therapy including intravitreal injections.
7. History of intraocular surgery in the past 3 months.
8. Anticipated cataract surgery in the next 6 months.
9. Any active infection or inflammation in the eye.
10. Cases where good quality imaging is not possible, either due to hazy media or extremely high myopia.
11. Patients with uncontrolled glaucoma, with IOP > 21mm Hg on 2 or more medications.
12. Patients with subfoveal scar or significant subretinal haemorrhage occupying more than 50% of lesion size.
13. Eyes with previous retinal detachment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 12 months
  Mean change in visual acuity from baseline to 54 weeks as measured by ETDRS chart

SECONDARY OUTCOMES:
Mean change in macular thickness on OCT from baseline to 54 weeks | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Raja Narayanan, MD, Principal Investigator — LV Prasad Eye Institute
Locations (1):
- LV Prasad Eye Institute, Hyderabad, Andhra Pradesh, India